CLINICAL TRIAL: NCT00023582
Title: HIV Prevalence, Incidence and HSV-2 Prevalence Among High-Risk MSM in Lima, Peru
Brief Title: HIV and Genital Herpes Among High-Risk Men Who Have Sex With Men (MSM) in Lima, Peru
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: HPTN 036
Record Dates: First submitted 2001-09-10; First posted 2001-09-11 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections; Herpes Genitalis; HIV Seronegativity; Syphilis
Keywords: Syphilis; Herpes Genitalis; Risk Factors; Incidence; Prevalence; Homosexuality, Male; Informed Consent; Peru; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Herpes Genitalis; Syphilis; Homosexuality, Male

SUMMARY:
The purpose of this study is to provide biomedical and behavioral information that is necessary for planning and starting HIV prevention trials in Lima, Peru.

The occurrence of HIV is high among men who have sex with men (MSM) in Lima, Peru, and bacterial sexually transmitted diseases (STDs) and HSV-2 (genital herpes) are very prevalent in HIV-positive and -negative MSM there. Methods to reduce both HIV and STDs are urgently needed among MSM in Peru. The information gained from this study is very important for future HIV prevention and vaccine trials that will take place in Peru.

DETAILED DESCRIPTION:
HIV incidence is high among MSM in Lima, Peru, and bacterial sexually transmitted diseases (STDs) and HSV-2 are prevalent in both recently and chronically HIV-infected MSM as well as HIV-uninfected MSM. Bisexual HIV-infected MSM could be an important "bridge" transmitting HIV and other STDs to women. Interventions to reduce both HIV and STDs are urgently needed among MSM in Peru. Given these associations and the high prevalence of STDs among MSM in Lima, prevention of HIV infections is dependent partially on innovative methods to control bacterial and viral STDs among high-risk HIV-uninfected MSM. The data from this prevention preparedness study is critical for future HIV prevention and vaccine trials that will be conducted in Peru.

All MSM are counseled and tested for HIV, HSV-2, and syphilis at the screening visit. [AS PER AMENDMENT 07/23/02: The syphilis test results are provided at screening, whereas the HIV and HSV-2 test results are provided at the enrollment visit.] High-risk HIV-uninfected MSM in Lima, Peru, are enrolled. Men are interviewed about risk behaviors in the past 6 months. Trained counselors provide risk-reduction counseling according to locally accepted standards. Men are followed at 3-month intervals for 1 year to determine the incidence of and risk factors for prevalent and incident HIV and HSV-2, and to evaluate the effectiveness of retention strategies. In the baseline questionnaire, 2 additional modules address sexual networks and willingness to participate in HIV vaccine or prevention trials, including an acyclovir trial. Study data are collected and entered into a local database.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for the initial screening visit if they are:

* Men aged 18 years and older who have had sex with another man in the past 12 months.

Volunteers may be eligible for enrollment if they:

* Are able to stay on the study for 12 months;
* Are willing and able to provide information on how they can be located;
* Have had high-risk sexual behavior and have tested negative for HIV.

Exclusion Criteria

Volunteers will not be eligible if they:

* Have obvious mental problems that would prevent them from fully understanding and participating in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, Study Chair
Locations (1):
- Rachael McClennen, Seattle, Washington, United States